CLINICAL TRIAL: NCT00431119
Title: A Comparison of Oral Methylprednisolone Plus Azathioprine or Mycophenolate Mofetil for the Treatment of Bullous Pemphigoid
Brief Title: Azathioprine or Mycophenolate Mofetil for Bullous Pemphigoid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beissert-BP#1
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2007-02-05 (Estimated); Status verified 2007-02

CONDITIONS: Bullous Pemphigoid
Keywords: bullous autoimmune disease; bullous pemphigoid; immunosuppressants; corticosteroids; mycophenolate mofetil
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Azathioprine; Mycophenolic Acid

INTERVENTIONS:
Drug: Azathioprine or Mycophenolate mofetil

SUMMARY:
To investigate the safety and efficacy of oral methylprednisolone combined with azathioprine or mycophenolate mofetil for the treatment of bullous pemphigoid.

DETAILED DESCRIPTION:
This multicenter randomized, non-blinded clinical trial compared two parallel groups of patients with bullous pemphigoid treated with oral methylprednisolone in combination with either azathioprine or mycophenolate mofetil. Patients were randomly assigned, irrespective of severity of disease, to receive either 0.5 mg per kg body weight (BW) methylprednisolone (Urbason®, Aventis Pharma, Bad Soden, Germany) with 2 mg per kg BW azathioprine sodium (Imurek®, GlaxoSmithKline, Munich, Germany) once daily or 0.5 mg per kg BW methylprednisolone once daily and 1,000 mg mycophenolate mofetil (CellCept® provided by Hoffmann-La Roche AG, Grenzach-Wyhlen, Germany), given twice daily (2 g/d). The initial dose was maintained until blister formation ceased, crusts as well as erosions disappeared, and re-epithelialization of previous lesions started. The corticosteroid dose was then sequentially reduced by 10 mg every two weeks until a dose of 20 mg per day was reached followed by a reduction in 5 mg-steps every two weeks until 10 mg per day. Afterwards, corticosteroid reduction was performed in 2.5 mg-steps every two weeks until zero. After discontinuation of corticosteroids azathioprine or mycophenolate mofetil doses were maintained at the initial dosage as monotherapy for an additional 4 weeks. Subsequently, azathioprine was reduced by 0.5 mg per kg BW every four weeks to a dose of 100 mg per day. Thereafter, azathioprine was tapered in 25 mg-steps every four weeks until discontinuation of treatment. Mycophenolate mofetil was reduced in 500 mg/d-steps every four weeks to 1,000 mg per day. From then on the mycophenolate mofetil dosage was decreased in 250 mg-steps every four weeks until discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical lesions suggestive of bullous pemphigoid
* subepidermal blistering upon histological analysis of skin biopsies
* linear deposition of IgG and C3 along the dermo-epidermal junction
* deposition of autoantibodies at the blister roof upon split-skin analysis

Exclusion Criteria:

* treatment with oral or topical corticosteroids, and other immunosuppressive drugs during the previous four weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 1997-10; Study Completion 2000-10

PRIMARY OUTCOMES:
The cumulative total methylprednisolone doses and rate of remission.

SECONDARY OUTCOMES:
Secondary outcome measures were safety profiles and duration of remission.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Beissert, MD, Principal Investigator — Dermatology, Univ. of Muenster, Germany
Locations (11):
- Germany (11):
  - Dermatology, Univ. of Cologne, Cologne
  - Dermatology, Univ. of Dresden, Dresden
  - Dermatology, Univ. of Duesseldorf, Düsseldorf
  - Dermatology, Univ. of Goettingen, Göttingen
  - Dermatology, Univ. Hospital Hannover, Hanover
  - Dermatology, Univ. of Kiel, Kiel
  - Dermatology, Univ. of Magdeburg, Magdeburg
  - Dermatology, Medical Faculty Mannheim, Univ. of Heidelberg, Mannheim
  - Dermatology, Municipal Hospital Minden, Minden
  - Dermatology, Univ. of Ulm, Ulm
  - Dermatology, Univ. of Wuerzburg, Würzburg

REFERENCES:
- [Background] Beissert S, Werfel T, Frieling U, Bohm M, Sticherling M, Stadler R, Zillikens D, Rzany B, Hunzelmann N, Meurer M, Gollnick H, Ruzicka T, Pillekamp H, Junghans V, Luger TA. A comparison of oral methylprednisolone plus azathioprine or mycophenolate mofetil for the treatment of pemphigus. Arch Dermatol. 2006 Nov;142(11):1447-54. doi: 10.1001/archderm.142.11.1447. PMID 17116835
- [Derived] Beissert S, Werfel T, Frieling U, Bohm M, Sticherling M, Stadler R, Zillikens D, Rzany B, Hunzelmann N, Meurer M, Gollnick H, Ruzicka T, Pillekamp H, Junghans V, Bonsmann G, Luger TA. A comparison of oral methylprednisolone plus azathioprine or mycophenolate mofetil for the treatment of bullous pemphigoid. Arch Dermatol. 2007 Dec;143(12):1536-42. doi: 10.1001/archderm.143.12.1536. PMID 18087004